CLINICAL TRIAL: NCT00980122
Title: Aggressiveness of Care at the End of Life in Cancer Patients
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Alvin Wong, National University Hospital, Singapore
Other Study IDs: MC05/30/07
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Advanced Cancer
Keywords: Advanced cancer patients dying in hospital receive aggressive cancer-specific therapy and supportive measures.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Cancer is the commonest cause of death in Singapore, and many cancer deaths occur in hospital.

Management of cancer patients is getting more complex with constant development of new drugs, interventional procedures and supportive measures. Despite this, the majority of advanced cancer patients will die from their disease or related complications.

There is a lack of data on the utilisation of health resources in advanced cancer patients in this country. In this study the investigators ask themselves how aggressive care was in the last 3 months of the patient's life. The investigators will be collecting data on specific cancer treatments, interventional procedures, and supportive measures.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer patients who passed away as an inpatient in NUH, under the department of Haematology Oncology.

Exclusion Criteria:

* Patients with haematologic malignancies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All advanced cancer patients who passed away in the National University Hospital during a defined 1 year period, will have a retrospective review of paper and electronic records.
  Study subjects are identified from the weekly mortality lists that are sent to the Department of Haemtology Oncology. We aim to include 250 patients in this retrospective study.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-03

PRIMARY OUTCOMES:
To describe the trends in the aggressiveness of care for advanced cancer patients near the end of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Braga S, Miranda A, Fonseca R, Passos-Coelho JL, Fernandes A, Costa JD, Moreira A. The aggressiveness of cancer care in the last three months of life: a retrospective single centre analysis. Psychooncology. 2007 Sep;16(9):863-8. doi: 10.1002/pon.1140. PMID 17245696
- [Background] Cintron A, Hamel MB, Davis RB, Burns RB, Phillips RS, McCarthy EP. Hospitalization of hospice patients with cancer. J Palliat Med. 2003 Oct;6(5):757-68. doi: 10.1089/109662103322515266. PMID 14622455